CLINICAL TRIAL: NCT03998540
Title: Improvement of DIAgnostic and Phenotype-genotype Correlation Studies in Patients With MYOpathy Suspected of TITinopathy
Acronym: DIAMYOTIT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0077; 2018-A02287-48 (Other: ANSM)
Record Dates: First submitted 2019-06-20; First posted 2019-06-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Myopathy; Phenotypic Abnormality; Genetic Disease
Keywords: titine; western blot
MeSH Terms: conditions — Muscular Diseases; Genetic Diseases, Inborn | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with myopathy suspected of titinopathy: Patients with myopathy in which one or more potentially pathogenic TTN variants have been previously identified (index cases and related cases affected). Muscle biopsy performed previously
  Interventions: Diagnostic Test: Western blot; Other: Protein interaction studies; Other: Mass Spectometry; Other: RNA seq

INTERVENTIONS:
Diagnostic Test: Western blot — Western-blot analysis of a giant protein, with specific antibodies directed against C-ter and N-Ter of the protein
Other: Protein interaction studies — Analyses of several interacting proteins by specific Western-blot and in-vitro tests.
Other: Mass Spectometry — samples previously used for western blotting will be subjected to mass spectrometry analysis
Other: RNA seq — analyze muscle gene expression in patients with titinopathies in our cohort by RNAseq

SUMMARY:
Due to the widespread use of NGS, TTN is emerging as a major causative gene in neuromuscular disorders, with high clinical heterogeneity. The mechanisms underlying the phenotypic variability and mode of inheritance (recessive or dominant) of titinopathies are poorly understood. They involve the primordial structural functions of titin on the formation and stability of the sarcomere, as well as its interactions with other proteins. We identified by NGS, in patients with skeletal myopathy (with or without cardiomyopathy), several potentially disease causing TTN variants. The specific aims of the present project are to implement functional studies (transcripts, protein analyses, in vitro protein-protein interaction studies) to evaluate the effect of TTN variants on the transcripts and protein in order to perform phenotype-genotype correlation studies. We participate to the national "titin network" and to international efforts for the understanding of the molecular bases of titinopathies. Genomic characterisation opens the way to develop cellular models of titinopathy, derived from patient biopsies. This is also a mandatory first step for the design of novel therapeutic approaches.

DETAILED DESCRIPTION:
Titinopathies are hereditary skeletal and cardiac myopathies due to alteration of titin, a giant elastic protein of the sarcomere. Due to the widespread use of next generation sequencing (NGS), the titin gene (TTN) is emerging as a major causative gene in neuromuscular disorders (NMDs), with high clinical and allelic heterogeneity. The mechanisms underlying the phenotypic variability and mode of inheritance recessive or dominant of titinopathies are poorly understood. They involve the primordial structural functions of the titin on the formation and stability of the sarcomere, as well as its interactions with other proteins. Effects of variants in TTN are variable, silent, recessive or dominant, and bioinformatics tools are not really efficient for interpretation of their functional impact, making them extremely difficult to interpret. Moreover, TTN variants are very frequent in the general population. Due to the huge size (3700kD) and complexity of titin, analyses of consequences of TTN variants on transcripts and protein are not performed commonly. There are few teams in the international community, but no team in France, that propose Western-blot (WB) analyses on titin as a diagnostic test. Moreover, this test allows to confirm the diagnosis only for recessive titinopathies due to truncating mutations, that are rare situations (<10% of suspected titinopathies). Concerning non-truncating variants, that are the most frequent ones (in particular missense variants), there are no functional diagnostic tests to assess their pathogenicity. Thus, expect the cases of recessive titinopathies due to compound heterozygous truncating mutations, it is not possible to confirm whether the phenotype of a patient is due to a titinopathy, leaving patients without diagnosis. It is thus important to implement functional tests to evaluate the pathogenic effects of TTN variants on titin abundance and functions.

This project comes from our NGS diagnostic results and will be the continuation of an ongoing AFM funded project (application 19958). We have identified by NGS, in patients with skeletal myopathy (with or without cardiomyopathy), several potentially disease causing TTN variants. Thanks to the AFM-funded project, we have analysed consequences of some TTN variants on splicing, and we are currently implementing experimental conditions to perform titin WB. In addition, we have observed that most non-truncating variants in TTN suspected to be pathogenic are located in titin domains interacting with myosin heavy-chain (MHC). In the hypothesis that they could have deleterious effects in the stability of interactions between titin and MHC in the sarcomere, we plan to implement functional tests to evaluate their consequences in titin-myosin interactions.

The specific aims of the present project will be to implement functional studies to evaluate the effect of TTN variants on the transcripts and protein in order to improve the diagnostic approach and to perform correlation studies with the modes of inheritance and the phenotypes. Innovative aspect of the project is the combination of several molecular and biochemical approaches on RNA (evaluation of the effects on transcription and/or splicing on titin transcripts in skeletal muscle of patients), protein (evaluation of the effects of all TTN variants on titin amount and size, by WB analyses on muscle biopsies) and protein-protein interactions (assessment of pathogenic impact of TTN variants located in titin-MHC interacting domains on interactions with MHC), that we will implement on the basis of technologies reported in academic research projects. The strength of our project is also based on our robust network with neurologists, neuro paediatricians, pathologists and other biological experts, within the organization in an interregional reference center of NMDs and in a national network of titinopathies, and the implication in the project of a neurologist (Dr Morales) through his PhD thesis, to carry out phenotype-genotype correlations studies.

Functional studies of the variants identified in the TTN gene should have strong impact for diagnosis of patients, that is important for its management and familial genetic counselling. The implemented tests will be available to the French network of titinopathies. This should solve the diagnosis of a large number of patients without clear diagnosis, and specify the frequency of involvement of titinopathies in myopathies. Improvement of diagnosis of titinopathies will have high socio-economic impacts because it will reduce the cost due to iterative diagnostic tests.

Phenotype-genotype correlation studies will allow expanding the mutation and clinical spectrum of titinopathies and participating to the international effort to understand the molecular bases of titinopathies, that is a mandatory first step to devise therapeutic approaches. In addition, genetic confirmation open the way to develop cellular models of titinopathy, derived from the tissues of patients. These models will be basis for proteomic and other functional studies to decipher the mechanisms of titinopaphies and to point to metabolic pathways that could be the target of pharmacological therapeutics.

For these reasons, the present application will constitute a major, original and innovative development to contribute to diagnosis and to the knowledge of molecular bases of titinopathies.

This study includes an ancillary study on the same cohort of patients and sample. The main objective is to evaluate the effects of TTN variants on the quantity and composition of titin peptides in patients' skeletal muscles.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed by a neurologist or a pediatric neurologist.
* Child or adult with congenital or progressive, proximal or distal myopathy
* Identification by NGS analysis of variant(s) in the potentially pathogenic TTN gene(s)
* Muscle biopsy performed previously
* Collection of the patient's (or one of his legal representatives if minor) non-opposition to participate in the present study and for the collection of the necessary biological material (muscle)
* Patient affiliated to or benefiting from a social security scheme

Exclusion Criteria:

* Absence of muscle sampling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with suspected titinopathy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of the relative quantity of titin protein | enrollment
  Evaluated by Western blot: normal or not, characterization of anomalies if any
Measurement of the relative size of titin protein | enrollment
  Evaluated by Western blot: normal or not, characterization of anomalies if any

SECONDARY OUTCOMES:
Measurement of consequences on interacting proteins | during 2 years
  Evaluation by Western blot: normal or not
Measurement of the consequences of TTN variants on titin transcripts | 2 years
  Evaluation by RT-PCR studies from muscle biopsies
Phenotype-genotype correlation studies | 2.5 years
  Correlation of clinicobiological data
Analyses of molecular bases of the different mode of inheritance of the disease | 2.5 years
  Integrated analyses of the complete biological data and correlation with the familial data
Mesurement of the level of interactions by in-vitro studies | during 2 years
  Evaluation by Western blot: normal or not
Evaluate the effects of TTN variants on the amount and composition of titin peptides in patient skeletal muscle | during 2 years
  By mass spectrometry
Evaluate the impact of TTN variants on titin expression and splicing in patient skeletal muscle | during 2 years
  using the poly-A tail selection protocol for mRNAs
Evaluate the impact of TTN variants on muscle gene expression levels by expression analysis of RNAseq data | during 2 years
  Expression analysis can be performed using R software and DESeq2 software.
Evaluate the effects of TTN variants on muscle protein partners. | during 2 years
  Quantitative proteomic analysis,mass spectrometry, will enable us to assess the quantity of muscle proteins, overall protein profile, in patients' muscle

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No